CLINICAL TRIAL: NCT06807502
Title: Evaluation of Circulating Tumor Cells (CTC) Relevance in Breast Cancer Follow-up Using the ScreenCell Device
Acronym: PROBE-CTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ScreenCell (Industry)
Collaborators: AXELYS SANTE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A01101-46
Record Dates: First submitted 2025-01-14; First posted 2025-02-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer, Metastatic; Breast Cancer Invasive; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: CTC; Circulating Tumor Cells; Detection; Breast Cancer; Follow-up; Liquid Biopsy; Blood Test
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplastic Cells, Circulating

STUDY DESIGN:
Intervention Model Description: Interventional study with minimal risk and constraints (RIPH2) comparative and open, non-randomized, on an in vitro diagnostic medical device.
  A case-control study with longitudinal, prospective, single-center follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Donor (Active Comparator): Participants with no history of cancer and free from any cancer at the time of inclusion
  Interventions: Device: The DM/DIV ScreenCell is the experimental product studied during this research
- Metastatic (Experimental): Participants with metastatic breast cancer or metastatic relapse of previously treated breast cancer with change of therapeutic line at the time of study inclusion
  Interventions: Device: The DM/DIV ScreenCell is the experimental product studied during this research
- No metastatic (Experimental): Participants with invasive breast cancer but non-metastatic
  Interventions: Device: The DM/DIV ScreenCell is the experimental product studied during this research

INTERVENTIONS:
Device: The DM/DIV ScreenCell is the experimental product studied during this research — The product is not used directly on the subject, but on a blood sample taken from the participant.

SUMMARY:
Liquid biopsy is a noninvasive method for detecting and quantifying circulating tumor cells (CTCs). Thanks to ScreenCell technology, this study aims to evaluate the evolution of the number of CTCs during breast cancer follow-up.

The identification and characterization of CTCs would make it possible to obtain information on the stage and molecular characteristics of cancer during follow-up

ELIGIBILITY:
INCLUSION CRITERIA

For all participants :

* Age greater than or equal to 18 years

For participants with metastatic breast cancer:

- Patient observed with metastatic breast cancer from the outset or metastatic fall from previously treated breast cancer with change of therapeutic line at the time of inclusion.

For participants with non-metastatic invasive breast cancer:

- Patient observed with non-metastatic infiltrative breast cancer who had not received any treatment at the time of inclusion (naïve to any treatment)

For healthy volunteers:

* Participant free of any cancer at the time of inclusion, confirmed using a mammogram whose results must be satisfactory, done at the latest one year before inclusion
* Participant with no history of cancer

EXCLUSION CRITERIA

For all participants:

* Age less than 18 years old
* Refusal to participate or withdrawal of consent
* Pregnant and/or breastfeeding women
* Discovery of a cancerous pathology (other than breast cancer for patients) during participant follow-up.

For participants with breast cancer:

- Absence of CTC during screening

For healthy volunteers:

* History of cancer
* Detection of CTC (positive profile) during screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as female are eligible to participate to evaluate breast cancer within a homogenized cohort, ensuring more relevant and reliable biostatistical analyses
Enrollment: 93 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of the kinetics of CTC during treatment | From enrollement to the end of follow up at 9 months
  Evolution of the number of CTC isolated by ScreenCell technology thanks to a blood draw during the therapeutic management of metastatic and infiltrative non-metastatic breast cancer patients. Average number of CTCs measured during the study (D0, W6, W12, W24, W36)

SECONDARY OUTCOMES:
Molecular characterisation of CTC | From enrollement to the end of follow up at 9 months
  Analysis of the expression of specific antigens and the presence of informative mutations on CTCs isolated by ScreenCell technology thanks to a blood draw during the therapeutic management of metastatic and infiltrative non-metastatic breast cancer patients during the study (D0, W6, W12, W24, W36)

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré Hartmann, Neuilly-sur-Seine, France